CLINICAL TRIAL: NCT02074475
Title: GE AOA Study Spin-off: Defining the Clinically Useful Range for Surgical Pleth Index
Brief Title: SPI Value Relevance in Clinical Practice
Acronym: SPIrelevance
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JH2013-1
Record Dates: First submitted 2013-12-19; First posted 2014-02-28 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Control group: The control group of three sites for larger Adequacy of Anaesthesia study. Total 150 patients
  Interventions: Other: Control group

INTERVENTIONS:
Other: Control group — A group of no Monitoring patients from larger AoA study with no adequacy of anaesthesia monitoring

SUMMARY:
Primary endpoint: Defining The optimal target range for Surgical Pleth index. Surgical Pleth Index (SPI, formerly used SSI = Surgical Stress Index) is a novel multivariate index, which is based on the sum of the normalized pulse beat interval (PBI) and the photoplethysmography. SPI indicates the balance between intensity of surgical stimulation and the level of anti-nociception (opioid analgesia and neural blockade). This study is a Spin off from a larger Adequacy of Anaesthesia study and aims on finding the most appropriate target range for SPI in order to avoid signs of inadequate anaesthesia. Patients are treated without monitoring adequacy of anaesthesia thus the values are collected blinded and analyzed afterwards in accordance of signs for inadequate anaesthesia. The study population will be 150 patients.

DETAILED DESCRIPTION:
Signs of non-adequate anaesthesia are motor and/or autonomic nervous system arousals during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent

  * Age 18-80 years of age
  * Surgery that is expected to last at least 2 hours under general anesthesia with endotracheal tube

Exclusion Criteria:

* Any subject that meets the definition of vulnerable subject as defined in ISO 14155:2011o Per ISO 14155:2011, a vulnerable subject is defined as an individual whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate

  * Any subject with a cardiac pacemaker
  * Any subject with atrial fibrillation at the time of obtaining the baseline values
  * Any subject with more than 5 ventricular extra systoles/minute at the time of obtaining the baseline values
  * Any subject who needs invasive blood pressure measurement
  * Any subject who show hemodynamics that would have qualified for being considered as a sign of inadequate anesthesia already at baseline:

    o Mean blood pressure below 60 mmHg or above 100 mmHg o HR below 45 /min or above 100/min
  * Any subject with epidural anesthesia or analgesia during the surgery. Epidural catheter may be placed pre-operatively, and used in the PACU, but not during the surgery
  * Any subject having surgery that requires prone position
* Any subject with very high body mass index (>35) because of incompatibility with the target controlled anesthesia models used

  * Any subject with known allergies to the specific anesthetic agents/ analgesic drugs intended for use in their surgeries
  * Any subject with laryngeal mask airway
  * Any subject who requires neuromuscular blocking agent infusion
  * Any subject who is going to have major surgery with a high risk of extensive blood loss
  * Any subject with known chronic use of opioids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients assessed for operation lasting more than two hours and requiring intubation.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
optimal maximum limit for SPI | 1 day
  SPI -value at a predefined criteria for signs of anaesthesia.

SECONDARY OUTCOMES:
Optimal lower limit for SPI | 1 day
  The measured lower limit SPI-value at the time point for signs of too deep anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jarkko Harju, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland